CLINICAL TRIAL: NCT01422694
Title: Studies on the Natural History and Pathogenesis of Spondyloarthritis
Brief Title: Natural History and Development of Spondyloarthritis
Status: Recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110223; 11-AR-0223
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Arthritis; Spondylitis, Ankylosing
Keywords: Sacroiliitis; Ankylosing Spondylitis; Spondyloarthritis; HLA-B27; Enthesitis-Related Arthritis; Natural History
MeSH Terms: conditions — Arthritis; Spondylitis, Ankylosing; Sacroiliitis; Spondylarthritis; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control: Healthy volunteers will be recruited to serve as controls
- Other Inflammatory Diseases: Subjects with Other Inflammatory Diseases
- Patients with Spondyloarthritis: Subjects with confirmed or probable SpA will be identified predominantly by physician referral.

SUMMARY:
Background:

- Spondyloarthritis (SpA) is a group of bone and joint disorders that may cause back and joint pain and stiffness. In some cases, SpA can lead to abnormal bone growth affecting the joints and spine. Some patients have SpA without ever developing these growths, while others develop them after only a few years. Researchers are interested in studying people with SpA and their relatives to determine which people are more likely to develop more severe conditions.

Objectives:

- To identify symptoms and medical tests that can help determine whether a person with SpA is at risk for developing more severe forms of the disease.

Eligibility:

* Individuals of any age who have been diagnosed with SpA.
* Healthy volunteer relatives (at least 6 years of age) of the individuals with SpA.

Design:

* Participants will be screened with medical records and family medical histories, and will be invited to the clinical center for the study.
* Participants with SpA will have a physical exam and medical history, including a study of joint movement, blood and urine tests, and questionnaires about pain and quality of life.
* Participants with SpA will have imaging studies, including magnetic resonance imaging (MRI). Other samples such as skin tissue and bone marrow may also be collected for study.
* Healthy volunteers will provide a blood sample and cheek cell samples.
* No treatment will be provided, although treatment options will be discussed....

DETAILED DESCRIPTION:
The purpose of this protocol is to study the natural history of spondyloarthritis (SpA) in children and adults. Spondyloarthritis encompasses a spectrum of immune-mediated inflammatory diseases that exhibit overlapping features, but differ from other types of inflammatory arthritis in genetic predisposition, pathogenesis, and outcome. Ankylosing spondylitis (AS), the most common form of SpA, frequently begins in an undifferentiated form with back pain and stiffness in adults, and leads to aberrant ossification and ankylosis (fusion) of the spine. In children, SpA rarely presents with back pain, but instead often begins with pain and stiffness in the hips and knees due to arthritis. Enthesitis, or inflammation where tendons and ligaments connect to bones, is more common in children. Our ability to recognize early forms of AS involving the axial skeleton, particularly in children, and our understanding of the cause and progression of this disease, is limited.

The goals of this natural history protocol are to establish a cohort of pediatric and adult patients with SpA to prospectively evaluate the signs and symptoms, magnetic resonance imaging (MRI) and X-ray findings, and bone and inflammatory biomarkers associated with axial disease. We will study pathogenic mechanisms including the role of AS susceptibility genes and their variants in causing disease, and will identify patients for possible entry into future treatment studies.

Patients enrolled in this protocol will undergo a history, physical examination, imaging studies, and laboratory evaluation. When clinically indicated, patients may also be evaluated for extra-articular manifestations such as acute anterior uveitis, psoriasis or other skin problems, and inflammatory bowel disease. Peripheral blood samples will be collected from affected patients, unrelated healthy volunteers, and in some cases unaffected family members to help identify and study the genes involved in SpA and their functions. We may ask some subjects to undergo skin biopsy or bone marrow aspiration for research purposes, or to provide a stool sample for analysis of microbiota. For some patients and family members, we may ask permission to perform whole genome or exome sequencing. Fibroblasts and/or peripheral blood cells obtained from patients will be induced to become pluripotent stem cells that can be maintained indefinitely in culture and differentiated into cell types that are relevant to pathogenesis. Successful completion of these studies will allow rheumatologists to better recognize early SpA with axial involvement, particularly in children, and will improve our understanding of disease pathogenesis.

ELIGIBILITY:
* INCLUSION CRITERIA

To be eligible for follow-up visits, patients must meet the Inclusion Criteria, but not the Exclusion Criteria. Subjects will provide informed consent and then be evaluated either in the outpatient or inpatient unit of the NIH Clinical Center.

* Subjects with known or suspected SpA.
* Family members of individuals with known or suspected SpA. Family members will not be asked to submit to bone marrow aspiration or interruption of therapy.
* Controls for clinical, cellular, molecular, and biochemical assays, and genetic evaluation will be enrolled. Individuals who undergo phlebotomy specifically to provide a control specimen will be 6 years of age or older, and not pregnant.
* Minor healthy volunteers undergoing imaging (SI and/or WB MRI) must be old enough to complete the procedure without sedation. Generally this requires that they be at least 6 years of age, so no healthy volunteers under age 6 will be enrolled.
* Pregnant people with SpA are allowed to enrolled. Pregnant people will not be asked to undergo an MRI and will not be asked to submit to skin biopsy or bone marrow aspiration.

EXCLUSION CRITERIA

* Inability to provide informed consent or, in the case of minors, unavailability of a parent or guardian.
* Presence of any medical condition that would, in the opinion of the investigators, confuse the interpretation of the study.
* Unavailability, or inability to comply with the schedule for follow-up visits.
* Children under the age of 2 years old.

The vast majority of minors with SpA or suspected SpA will be 6 years of age or older. However, it is possible that children younger than age 6 will be evaluated. If children under age 6 are referred for evaluation, we will ensure that they do not have any acute or chronic comorbidity that would preclude them from being safely evaluated at the NIH Clinical Center. Such patients would be referred to other appropriate pediatric hospitals.

Based on estimates of the incidence and prevalence of SpA in the pediatric and adult populations we set the accrual ceiling up to 2000. We hope to enroll up to 100 patients per year.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with spondyloarthropathies.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-08-12 (Actual)

PRIMARY OUTCOMES:
Progression from SpA to Axial Spa and to AS | 10 years
  sacroiliac damage on x-ray

SECONDARY OUTCOMES:
Measures of disease activity (BASDAI and ASDAS) and function (BASFI). | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Lotfi-Emran, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-AR-0223.html